CLINICAL TRIAL: NCT01437592
Title: A Trial Investigating the Pharmacokinetic Properties of NN1250 in Healthy Chinese Subjects
Brief Title: Investigating the Pharmacokinetic Properties of NN1250 in Healthy Chinese Subjects
Status: Completed | Phase: Phase 1 | Type: Interventional
Sponsor: Novo Nordisk A/S (Industry)
Responsible Party: Sponsor
Allocation: Non-Randomized | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: NN1250-1999; U1111-1122-6475 (Other: WHO)
Record Dates: First submitted 2011-09-09; First posted 2011-09-21 (Estimated); Last update posted 2019-05-30 (Actual); Status verified 2019-05

CONDITIONS: Diabetes; Healthy
MeSH Terms: conditions — Diabetes Mellitus | interventions — insulin degludec

STUDY DESIGN:
Oversight: Data Monitoring Committee: No

ARMS (1):
- IDeg (Experimental)
  Interventions: Drug: insulin degludec

INTERVENTIONS:
Drug: insulin degludec — For each subject, a single dose of NN1250 will be administered subcutaneously (under the skin)

SUMMARY:
This trial was conducted in Asia. The aim of this trial was to investigate the pharmacokinetic properties (the effect of the investigated drug on the body) of NN1250 (insulin degludec) in healthy Chinese subjects.

ELIGIBILITY:
Inclusion Criteria:

* Male or female Chinese subject aged 18-45 years (both inclusive)
* Considered generally healthy upon completion of medical history, physical examination, vital signs and electrocardiogram (ECG), as judged by the Investigator
* Body mass index 19.0-24.0 kg/m^2 (both inclusive)

Exclusion Criteria:

* A history of any illness that, in the opinion of the Investigator, might confound the results of the trial or pose risk in administering the trial product to the subject
* Subject who has donated any blood or plasma in the past month or more than 400 mL within 3 months prior to screening
* Not able or willing to refrain from smoking during the inpatient period

Ages: 18 Years to 45 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult
Enrollment: 24 (Actual)
Dates: Start 2011-09-06 (Actual); Primary Completion 2011-11-22 (Actual); Study Completion 2011-11-22 (Actual)

PRIMARY OUTCOMES:
Area under the serum insulin degludec concentration-time curve | From 0 to 120 hours after single dose

SECONDARY OUTCOMES:
Maximum observed serum insulin degludec concentration | 0-24 hours (derived on treatment day 1).
Time to maximum observed serum insulin degludec concentration | 0-24 hours (derived on treatment day 1).

CONTACTS AND LOCATIONS:
Overall Officials: Global Clinical Registry (GCR, 1452), Study Director — Novo Nordisk A/S
Locations (1):
- Novo Nordisk Investigational Site, Beijing, Beijing Municipality, China

REFERENCES:
- [Background] Pei H, Jiang J, Bardtrum L, Haahr H. Pharmacokinetic properties of insulin degludec in healthy Chinese subjects. Diabetes Manag 2019;9(1):20-7
- See also: Clinical Trials at Novo Nordisk — http://novonordisk-trials.com